CLINICAL TRIAL: NCT07341802
Title: Pilot Feasibility Study of a Fall Prevention Exercise Programme for Community-dwelling Older Adults in Nanchang, China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UM.TNC2/UMREC_3210
Record Dates: First submitted 2025-12-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Fall Prevention
Keywords: Fall prevention; Exercise adherence; Older adults
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In addition to outcomes assessors, the data analysts are masked to group allocation. The dataset provided for analysis uses coded group labels ("Group A" and "Group B"), and the analysts remain blinded until after the primary analyses are complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe & Joyful Walk (Experimental): Participants will attend 24 instructor-led group sessions over 12 weeks, focusing on balance, strength, and functional exercises. In addition, they will complete unsupervised home-based practices so that, together with the group sessions, they achieve the weekly target of 120 minutes of exercise. Instructional videos, printed manuals, and WeChat reminders will support independent practice.
  Interventions: Behavioral: Safe & Joyful Walk
- Tai Chi (Active Comparator): Participants will attend 24 instructor-led group sessions over 12 weeks, practicing 24-form simplified Yang-style Tai Chi. In addition, they will complete unsupervised home-based practices so that, together with the group sessions, they achieve the weekly target of 120 minutes of exercise. Instructional videos, printed manuals, and WeChat reminders will support independent practice.
  Interventions: Behavioral: Tai Chi

INTERVENTIONS:
Behavioral: Safe & Joyful Walk — A 12-week group-based exercise programme designed to improve balance, strength, and functional mobility. Participants attend 24 instructor-led sessions and complete additional home-based practices, with the combined duration of group and home sessions reaching the target of 120 minutes of exercise per week. Instructional videos, printed manuals, and WeChat reminders support adherence.
  Arms: Safe & Joyful Walk
Behavioral: Tai Chi — A 12-week group-based Tai Chi programme using the simplified 24-form Yang-style routine. Participants attend 24 instructor-led sessions and complete additional home-based practices, with the combined duration of group and home sessions reaching the target of 120 minutes of exercise per week. Instructional videos, printed manuals, and WeChat reminders support adherence.
  Arms: Tai Chi

SUMMARY:
The goal of this pilot clinical trial is to evaluate the feasibility of a fall prevention exercise programme for older adults living in urban communities in China. The study will also gather preliminary data on whether the programme can improve adherence to exercise and reduce falls.

The main questions it aims to answer are:

* Is the Safe & Joyful Walk programme feasible and acceptable for older adults in urban China?
* Does the programme help participants stick to regular exercise?
* Does the programme show early signs of improving balance, walking speed, and reducing falls?

Researchers will compare the Safe & Joyful Walk programme to Tai Chi to see which approach may better support exercise adherence and fall prevention.

Participants will:

* Attend 24 instructor-led group exercise sessions over 12 weeks
* Complete additional unsupervised home-based exercise practices during the same 12-week intervention period
* Continue unsupervised exercises during a 24-week follow-up period to assess long-term adherence
* Complete surveys, interviews, and physical tests at baseline, 12 weeks, and 36 weeks
* Record their exercise and any falls in diaries and calendars

ELIGIBILITY:
Inclusion Criteria:

* age 60 years or older;
* Mandarin-speaking;
* independent in activities of daily living;
* able to walk 10 m without the use of a walking aid;
* willingness to provide informed consent and comply with the study protocol.

Exclusion Criteria:

* an acute psychiatric condition with psychosis;
* an unstable medical condition that would preclude safe participation;
* a progressive neurological condition (such as Parkinson's disease, multiple sclerosis, Meniere's disease);
* cognitive impairment defined as a Pfeiffer Short Portable Mental Status Questionnaire (SPMSQ) score <8 ;
* residing in residential aged care, currently participating in a fall prevention trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety of the intervention (adverse events) | Baseline to 36 weeks.
  Safety will be assessed by the number and type of adverse events reported by participants and recorded in exercise diaries throughout the 12-week programme and 24-week follow-up.
Recruitment rate | Up to 4 weeks
  Recruitment will be assessed by the proportion of eligible participants enrolled, recorded in the Study Screening Log.
Attrition rate | Baseline to 36 weeks
  Attrition will be assessed by the proportion of participants who withdraw before completing the 36-week follow-up, recorded in the Withdrawal Log.
Fall rate | Baseline to 36 weeks
  Falls will be tracked using participant fall calendars with monthly telephone verification; outcomes include number of falls and fallers over the 36-week period.

SECONDARY OUTCOMES:
Attendance at group sessions | Baseline to 12 weeks
  Attendance will be assessed by the number and proportion of sessions attended, recorded in Attendance Logs.
Adherence to home-based practice | Baseline to 36 weeks
  Adherence will be assessed using Exercise Diaries, documenting frequency and duration of home-based practice.
Balance confidence (Activity-specific Balance Confidence Scale, ABC) | Baseline, 12 weeks and 36 weks
  Balance confidence will be assessed using the Activity-specific Balance Confidence (ABC) Scale, a 16-item self-report questionnaire measuring confidence in performing daily activities without losing balance. Scores range from 0% to 100%, with higher scores indicating greater balance confidence.
Gait speed (4-meter gait speed test) | Baseline, 12 weeks and 36 weeks.
  Usual gait speed will be measured over 4 meters using standardized procedures; faster speed indicates better performance.
Balance performance (One-Leg Stance test) | Baseline, 12 weeks and 36 weeks.
  Static balance will be assessed using the One-Leg Stance test; longer stance time indicates better balance.

OTHER OUTCOMES:
Socio-demographic and clinical characteristics | Baseline
  Socio-demographic and clinical characteristics-including age, sex, education level, and 12-month fall history-will be collected using the Demographic Information and Fall History Form. These variables will be summarized using descriptive statistics (e.g., means and standard deviations for continuous variables; frequencies and percentages for categorical variables) to describe the study sample.
Programme acceptability | Week 12 and week 36
  Programme acceptability will be assessed using a structured questionnaire and semi-structured interviews. The questionnaire consists of five yes/no items addressing satisfaction, perceived benefits, interest, fatigue, and willingness to continue the programme. Quantitative acceptability will be determined by calculating the proportion of affirmative ("Yes") responses; if at least 50% of the responses are affirmative, the programme will be considered acceptable. Qualitative acceptability will be explored through semi-structured interviews to capture participants' experiences, perceived benefits, and barriers to participation.

CONTACTS AND LOCATIONS:
Locations (1):
- QingShanHu University for the Elderly, Nanchang, Jiangxi, China